CLINICAL TRIAL: NCT01559987
Title: A Randomized Parallel Method Development Study Comparing Clinical to Subclinical Effects From Oral Cleaning Modalities
Brief Title: Dental Plaque Removal Study
Acronym: PAU2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Philips Oral Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MAH-11-0059
Record Dates: First submitted 2012-03-06; First posted 2012-03-21 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2017-01

CONDITIONS: Gingivitis; Gum Disease
Keywords: plaque removal methods; oral hygiene devices
MeSH Terms: conditions — Gingivitis; Gingival Diseases

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Other): ADA (American Dental Association) Reference Manual Toothbrush (MTB)
  Interventions: Other: Manual Toothbrush only
- Test (Other): MTB + Floss
  Interventions: Other: MTB + Floss (MTB+Floss)
- MTB + Waterpik Ultra Water Flosser High (Experimental): MTB + Waterpik Ultra Water Flosser High
  Interventions: Other: MTB + Waterpik Ultra Water Flosser 'High'

INTERVENTIONS:
Other: Manual Toothbrush only — ADA (American Dental Association) Reference Manual Toothbrush (MTB)
  Arms: Control
Other: MTB + Waterpik Ultra Water Flosser 'High' — MTB + Waterpik Ultra Water Flosser 'High'
  Arms: MTB + Waterpik Ultra Water Flosser High
Other: MTB + Floss (MTB+Floss) — MTB + Floss (MTB+Floss)
  Arms: Test

SUMMARY:
The purpose of this research study is to investigate water flow in dental devices and to understand the function of water flow behind oral hygiene improvements. Understanding this mechanism may help with the design of future products.

DETAILED DESCRIPTION:
The overall clinical response (plaque, gingivitis, bleeding) in participants with varying stages of gingival health as well as the causative or indicative hallmarks of selected biological responses underpinning the overt clinical manifestations described above will be evaluated. The chief biological response that will be investigated is how a reduction in the concentration of bacterial lipopolysaccharide endotoxins (LPS) in interproximal plaque may influence improvements in the clinical response (e.g., through mitigation of bleeding) when compared to a change in the plaque biomass within which a large component of the endotoxins reside. The hypothesis is that improvements in clinical bleeding may result more from the removal or reduction of toxic bacterial products that serve as the direct impetus of the inflammatory response rather than from sheer bulk removal of interproximal plaque. From a methods development perspective, this study will also assess the feasibility of measuring endotoxin load from clinical samples. Ultimately it is anticipated that a comprehensive evaluation of clinical benefits conferred by continuous fluid streaming will emerge upon analysis of the relationships between clinical and biological data sets, particularly where causal relationships may exist between both parameters.

The devices used in this study are subject only to Class I (general controls) and considered exempt from the premarket notification procedures and not subject to section 510(k), 515, or 520(m,) of the FDC Act in order to be legally marketed. Thus, the study does not meet the definition of an Applicable Clinical Trial.

ELIGIBILITY:
Inclusion Criteria:

* are in good general health
* are 18 - 75 years old;
* have and will abstain from all oral care in the 12 hours prior to each scheduled appointment, but no more than 18 hours prior.
* have and will abstain from consumption of apples and other sticky fruits in the 12 hours prior to each appointment.
* agree to abstain from eating, drinking, chewing gum, and the use of breath mints, etc in the one hour preceding saliva collection at Visits 2 and 3
* have a minimum of 20 natural teeth (excluding 3rd molars);
* have 2 qualifying Interproximal Unit test sites in each posterior quadrant from 3 approximating teeth (see Section 5.1.1, Interproximal Unit (IU)Test Site Selection, for definition);
* present with one of the following three categories:
* BGI-gingivitis: all PD<3mm, BOP>10%;
* BGI-periodontitis (P2): 1+ site with PD>3mm, BOP>10% but <50%
* BGI-periodontitis (P3): 1+ site with PD>3mm, BOP>50%
* have provided written informed consent and are willing to participate and be available at all times required for participation
* are willing and able to fully understand and comply with the written and verbal study instructions provided in English
* agree to return all study materials at the final visit

Exclusion Criteria:

* have systemic diseases, Down's syndrome, or known AIDS/HIV;
* have Diabetes
* are a smoker
* are pregnant or nursing by participant report;
* have a cardiac pacemaker or AICD
* are undergoing or require extensive dental or orthodontic treatment;
* have had oral or gum surgery in the previous 2 months;
* require antibiotic treatment for dental appointments;
* have used antibiotics within 4 weeks of enrollment
* are currently using prescription-dose anti-inflammatory medications or anticoagulants (including aspirin)
* have heavy deposits of calculus, either supragingival and/or subgingival;
* have extensive crown or bridge work and/or rampant decay;
* currently use bleaching trays;
* have any oral or extraoral piercing on lips or in mouth with ornament or accessory;
* have a professional prophylaxis within 4 weeks of study;
* have participated in a prior study ≤ 20 days;
* participated in Philips study DRC-0742;
* are employed by an oral healthcare products company or dental research institution (i.e., dental school: administrative staff, assistants, hygienists, and research students).
* are a dentist, dental student or dental professional

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
residual protein concentration in posterior sites following in-clinic use of MTB (Manual Toothbrush)+Waterpik Ultra Waterflosser 'high', MTB+floss or MTB alone | Baseline and Week 2
  The primary endpoint of this study is the residual protein concentration in posterior sites following in-clinic use of MTB+Waterpik Ultra Waterflosser 'high', MTB+floss or MTB alone.

SECONDARY OUTCOMES:
Modified Gingival Index, Gingival Bleeding index, Plaque Index, and clinical attachment level). | Baseline and Week 2
  To evaluate the impact of a fluid cleaning principle (MTB+Waterpik Waterflosser) relative to MTB+Floss and MTB alone on clinical outcomes: Modified Gingival Index, Gingival Bleeding index, Plaque Index, and clinical attachment level.
Number of Adverse Events and Intraoral Exams | Baseline and week 2
  Safety endpoints based on adverse event reports and intraoral exam (soft tissue evaluation)findings.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Offenbacher, DDS, PhD, MMSc, Principal Investigator — UNC School of Dentistry
Locations (1):
- General and Oral Health Center, Chapel Hill, North Carolina, United States